CLINICAL TRIAL: NCT07178223
Title: TRACE - A Single Arm Trial of Thumb Base Replacement Arthroplasty for Osteoarthritis Compared to External Controls
Brief Title: TRACE - Thumb Base Replacement Arthroplasty for Osteoarthritis.
Acronym: TRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Wilcke, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thumb base arthroplasty
Record Dates: First submitted 2025-08-30; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis of the CMC-1 Joint
Keywords: cmc-1; osteoarthritis; thumb base; Arthroplasty; prosthesis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Single arm with external control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroplasty (Other): Arthroplasty CMC-1
  Interventions: Procedure: Arthroplasty CMC-1

INTERVENTIONS:
Procedure: Arthroplasty CMC-1 — Touch Touch® dual-mobility Arthroplasty CMC-1 joint (Kerimed). Dorsal approach. Conical cup. Soft dressing 3 weeks. Loading allowed after 2 months.

SUMMARY:
Osteoarthritis in the base of the thumb is one of the most common forms of hand arthritis. It usually appears in middle age, particularly in women, and can cause significant pain and loss of function. Early treatment often includes splints, painkillers, joint protection techniques, or steroid injections. If these measures are not enough, surgery is considered.

The current standard operation in Sweden is trapeziectomy-removing the trapezium. This usually gives good pain relief at rest, but many patients continue to experience pain when loading the hand and reduced grip strength. Another surgical option is trapeziometacarpal limited excision (TLE), where only part of the bone is removed to keep the thumb slightly longer, which may improve strength. Both procedures are non-implant surgeries.

A newer alternative is total joint arthroplasty (TJA), where the joint is replaced with a prosthesis. Early studies suggest that this may allow for quicker recovery and possibly better strength compared to trapeziectomy. However, it is more expensive and carries higher risks, such as implant loosening or dislocation. So far, research has not proven that it offers better long-term results.

The TRACE study (A single arm trial of Thumb base Replacement Arthroplasty for osteoarthritis Compared to External controls) is designed to help answer this question. Instead of randomizing patients, this study will follow a group of people receiving thumb joint replacement and compare them to an existing group of patients who already took part in a randomized trial of trapeziectomy and TLE. This design allows the researchers to study results more quickly and with fewer resources, while still ensuring meaningful comparisons.

The main research question of this study is whether joint replacement gives better pain relief when loading the thumb 10 years after surgery compared to traditional non-implant operations in patients with painful thumb base osteoarthritis. Secondary questions include whether joint replacement improves patient-reported outcomes, hand function, and strength, and whether it leads to more or fewer complications at 1, 3, and 5 years after surgery.

90 patients will be included in the replacement group, using a dual mobility prosthesis. Their outcomes will be compared with 90 patients from the earlier trial (45 trapeziectomy and 45 limited trapeziometacarpal joint resection - TLE). The study will track pain, daily hand function, strength, range of motion, and complications such as infection or the need for further surgery. Data will be collected regularly for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis in the thumb base. Radiological Eaton class 1-3 (Ladd et al. 2015).
* Clinical signs of thumb base osteoarthritis: pain at palpation of the CMC-1 joint and pain during provocation/grinding test.

The inclusion criteria are identical to those of the control population.

Exclusion Criteria:

* Rheumatoid arthritis.
* Ongoing infection in the hand or wrist.
* History of gout or pseudogout in the hand.
* Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).
* Chronic pain syndrome / centralized pain.
* Intra-articular corticosteroid injection in the affected joint within 3 months. -Eaton Littler class 4 (symptomatic STT joint osteoarthritis).

The previously described exclusion criteria are identical to those of the control population. In addition patients with severe deformation of the trapezium, to the extent that it is not possible to place a prosthetic cup, will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain on load in the thumb 10 years postoperatively. | 10 years postoperatively
  Pain on load is rated with a self-administered 11-point numerical rating scale (NRS) 0-100 from the HQ-7 questionnaire. Higher score means more pain. The participants are asked to rate the pain the previous week.

SECONDARY OUTCOMES:
Pain on load in the thumb 3 and 6 months, 1, 3, and 5 years postoperatively. | from enrollment to 5 years postoperatively
  Pain on load is rated with a self-administered 11-point numerical rating scale (NRS) 0-100 from the HQ-7 questionnaire. Higher score means mote pain. The participants are asked to rate the pain the previous week.
HQ-8 score 3 and 6 months, 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively
  Self-administered 11-point numerical rating scale (NRS) 0-100 symptoms questionnaire. Symptoms inlcude pain at rest, pain on motion, stiffness, weakness. Higher score means more symptoms. HQ-8 is the symptom-rating scale in the Swedish Hand surgical quality registry (HAKIR).
Patient-rated Wrist and Hand (PRWHE) score 3 and 6 months, 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively
  Patient-rated Wrist and Hand (PRWHE). Scale 0-100, higher score means more pain and disability,
Distability of the Arm, Hand and Shoulder (DASH) score 3 and 6 months, 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively.
  Distability of the Arm, Hand and Shoulder (DASH) score range from 0 to 100, higher score means more disability,
Thumb range of motion 3 and 6 months, 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively
  Palmar and radial abduction (degrees) of the first metacarpal measured with a goniometer
Adverse events | From enrollment to 10 years postoperatively.
  Number of particiant with a diagnosed infection, complex regional pain syndrome (CRPS), superficial radial sensory nerve injury or revision surgery required.
Thumb strength 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively
  Key pinch and three-finger pinch measured with a pinch gauge (kilograms).
Hand strength 1,3, 5 and 10 years postoperatively | From enrollment to 10 years postoperatively
  Full hand grip strength measured with Jamar (kilograms).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilcke, Associate professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Handkirurgiska kliniken Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
A description of the variables collected throughout the trial and used in the results publication will be provided when the study is finished.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 6 years after the publication of the final (10 years) results.
Access Criteria: Data will be shared for systematic reviews/metananalyses. The statistical methods for those analyses need not to be approved by an independent review.
  A proposal that describes planned analyses must be submitted by e-mail to the corresponding author who will review requests for IPD sharing.